CLINICAL TRIAL: NCT00220805
Title: Multicenter, Randomized, Double-blind, Placebo-controlled, Study to Evaluate the Efficacy and Safety of IGIV-C, 10% Treatment in Subjects With Pure Occult Choroidal Neovascularization Due to Age Related Macular Degeneration
Brief Title: Use of Immune Globulin Intravenous (Human) To Treat Age-Related Macular Degeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 100586
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Results first posted 2016-03-21 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-02

CONDITIONS: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — gamma-Globulins; Caprylates; Immunoglobulins, Intravenous; Albumins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental)
  Interventions: Drug: Immune Globulin Intravenous [Human], 10% Caprylate/Chromatography Purified
- Group 2 (Placebo Comparator)
  Interventions: Drug: Albumin (Human) 25%, United States Pharmacopeia (USP)

INTERVENTIONS:
Drug: Immune Globulin Intravenous [Human], 10% Caprylate/Chromatography Purified — The dose per infusion cycle was 2 g/kg body weight over 5 consecutive days (= 4 mL/kg body weight/infusion). The infusion duration was approximately 1.5 - 2 h.
  Other Names: Gamunex®; IGIVnex®; Gaminex; IGIV-C; IGIV-C, 10%; Immune Globulin IV (Human), 10% (IGIV); Immune Globulin IV (Human), 10% by Chromatography Process; IGIV; IVIG; BAY 41-1000; TAL-05-00004; NDC 13533-645-12; NDC 13533-645-15; NDC 13533-645-20; NDC 13533-645-24; NDC 13533-645-71
  Arms: Group 1
Drug: Albumin (Human) 25%, United States Pharmacopeia (USP) — Albumin (Human) 20% or 25% will be diluted with 5% glucose to a final concentration of 0.1%.
  Other Names: Plasbumin®-20; Plasbumin®-25; Plasbumin®-20 (Low Aluminum); Plasbumin®-25 (Low Aluminum); Albumin (Human) 20%, USP; TAL-05-00007; TAL-05-00008; TAL-05-00024; TAL-05-00025; BAY 34-9255; NDC 13533-683-20; NDC 13533-683-71; NDC 13533-684-16; NDC 13533-684-20; NDC 13533-684-71; NDC 13533-691-20; NDC 13533-691-71; NDC 13533-692-16; NDC 13533-692-20; NDC 13533-692-71
  Arms: Group 2

SUMMARY:
This study will evaluate visual improvement in patients treated with Immune Globulin Intravenous (Human), 10% Caprylate/Chromatography Purified (IGIV-C) or placebo who have Age-Related Macular Degeneration (AMD) with occult Choroidal Neovascularization (CNV).

DETAILED DESCRIPTION:
The purpose of this trial is to investigate the effect of IGIV-C in subjects suffering from AMD with occult CNV where fewer treatment options exist for patients with this disease form.

This study is designed as a randomized, double-blind, parallel group, placebo-controlled prospective trial. Sixty patients, 30 per treatment group, with newly diagnosed pure occult CNV defined by angiography diagnostic criteria will be enrolled. If a subject has more than one eye affected with occult CNV, the eye with the better vision as measured by visual acuity ( Logarithm of the Minimum Angle of Resolution [LogMAR] score) will be entered as the study eye.

Patients will be randomized to receive either IGIV-C at a dose of 2 g/kg body weight (bw) over 5 consecutive days or matching placebo. Additional 2 study drug treatment courses (IGIV-C or matching placebo) will be administered every 4 weeks at the same dose of 2 g/kg bw given over 5 days. Subjects' visual acuity will be measured and reported as LogMAR at screening, week 0 (baseline), day 5, week 4, week 8 and week 12. If at anytime during the study the subject's visual acuity worsens by ≥ 2 lines (0.2 on the LogMAR score), then a slit lamp examination will be performed and an angiogram will be conducted; the patient would be discontinued if the worsening is due to some other reason outside of the occult CNV or if the disease has changed from pure occult to the classic or mixed form.

Subjects will be evaluated for efficacy (LogMAR score) at endpoint (at week 12 or at last LogMAR assessment at or after week 8, if the subject prematurely discontinues the trial).

At the end of the treatment period (week 12), patients will be entered into a 3 month observation period with monthly visual acuity LogMAR score assessments.

ELIGIBILITY:
Inclusion Criteria:

* The best corrected visual acuity must be in the range of 20/40 to 20/200 on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart (0.5 - 0.1).
* Patient complaint of visual loss within the last three months prior to study entry.
* Documented visual loss on a visual acuity chart in the 3-month period prior to the beginning of the run-in period.
* Signed written informed consent prior to initiation of any study-related procedures.

Exclusion Criteria:

* Treatment with IGIV within the last 3 months prior to the run-in.
* Previous photodynamic therapy (PDT) or vitrectomy or transpupillary thermotherapy (TTT) or any specific pre-treatment of CNV
* Subfoveal blood in the study eye if ≥ 1/2 disc diameter as measured by slit lamp during run-in period.
* History of anaphylaxis or severe systemic response to immunoglobulin or with a blood product.
* Cardiac insufficiency (NYHA III/IV), cardiomyopathy, significant cardiac dysrhythmia requiring treatment, unstable or advanced ischemic heart disease, or severe or uncontrolled hypertension (diastolic > 95 mmHg or systolic >170 mmHg)
* Females, who are pregnant, breast feeding, or if of childbearing potential, unwilling to practice adequate contraception throughout the study.
* History of renal insufficiency or serum creatinine levels > 221 µmol/L (2.5 mg/dL).
* Known selective immunoglobulin A (IgA) deficiency
* Other investigational drugs received within the past 3 months.
* Conditions whose symptoms and effects could alter protein catabolism and/or immunoglobulin (IgG) utilization (e.g. protein-losing enteropathies, nephrotic syndrome).
* Known hypercoagulable state.
* Patients on continuous systemic steroid treatment
* Mentally challenged adult subjects who cannot give independent informed consent.
* History of thromboembolic events.
* Diabetes mellitus requiring drug treatment.
* Known severe hypersensitivity to sodium fluorescein.
* Acute or known ocular diseases such as glaucoma, arterial or venous occlusions, acute ischemic optic-neuropathy, impairment of visual acuity due to opacities in the lens (LOCSIII: NO 5-6 or C: 4-5 or P 4-5) or vitreous which may influence the evaluation of the therapeutic effect.

Min Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2004-01; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brunner, MD, Principal Investigator — Center of Ophthalmology, University of Cologne, Germany
Locations (7):
- Germany (7):
  - Universitatsklinikum Aachen, Augenklinik, Aachen
  - Medizinische Einrichtungen der Universitat zu Koln, Centrum fur Augenheilkunde, Cologne
  - Augenklinik Tausendfensterhaus, Duisburg
  - St. Martinus-Krankenhaus, Augenabteilung, Düsseldorf
  - Medizinische Eirnrichtungen der Universitat Essen, Klinik fur Erkrankungen des hinteren Augenabschnittes, Essen
  - Kliniken und Polikliniken der Albert Ludwigs Universität, Freiburg im Breisgau
  - Klininkum der Eberhard-Karls-Universitat Tubingen, Universitats-Augenklinik, Tübingen

REFERENCES:
- See also: FDA Approved Product Labeling Information - Gamunex® — http://www.talecris-pi.info/inserts/gamunex.pdf
- See also: FDA Approved Product Labeling Information - Plasbumin®-20 (Low Aluminum) — http://www.talecris-pi.info/inserts/plasbumin20la.pdf
- See also: FDA Product Approval — http://www.fda.gov/BiologicsBloodVaccines/BloodBloodProducts/ApprovedProducts/LicensedProductsBLAs/FractionatedPlasmaProducts/ucm089390.htm
- See also: FDA Approved Product Labeling Information - Plasbumin®-25 (Low Aluminum) — http://www.talecris-pi.info/inserts/plasbumin25la.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 96 subjects were enrolled (signed the informed consent and screened) in this study at 6 German study centers.
Pre-assignment Details: Of the 96 enrolled subjects, 14 subjects withdrew their consent for participation before randomization and an additional 25 subjects were withdrawn before randomization because of violations of inclusion/exclusion criteria or because their angiograms were rejected by the central reading site as not meeting the pre-specified criteria.
Groups:
- IGIV-C 10%: Immune Globulin Intravenous [Human], 10% Caprylate/Chromatography Purified
- Placebo: Albumin (Human) 25%, United States Pharmacopeia (USP)
Period: Overall Study
Arm/Group | IGIV-C 10% | Placebo
Started | 30 | 27
Completed | 22 | 16
Not Completed | 8 | 11
Not completed — Adverse Event | 1 | 3
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Develop. of choroidal neovascularization | 3 | 8

BASELINE CHARACTERISTICS:
Population: The intent to treat (ITT) population, which was defined as the primary analysis population, comprised 29 subjects treated with IGIV-C 10% and 24 subjects treated with placebo. A total of 4 subjects were excluded from the ITT population: 1 from IGIV-C 10% and 3 from Placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | IGIV-C 10% | Placebo | Total
Number analyzed (Participants) | 29 | 24 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 25 | 20 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.724 (8.417) | 74.042 (10.217) | 74.415 (9.189)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 37
  Male | 9 | 7 | 16
Region of Enrollment [Number; unit: participants]
  Germany | 29 | 24 | 53
Visual Acuity Score (VAS) of the Study Eyes [Mean (Standard Deviation); unit: units on a scale] | 55.9 (10.4) | 58.4 (7.7) | 57.0 (9.3)
Logarithm of the Minimum Angle of Resolution (LogMAR) of the Study Eyes [Mean (Standard Deviation); unit: LogMAR] | 0.581 (0.209) | 0.533 (0.153) | 0.559 (0.186)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Visual Acuity (Logarithm of the Minimum Angle of Resolution [LogMAR]) Score From Baseline for IGIV-C, 10% Compared to Placebo at Week 12 or at Last LogMAR Assessment (Conducted at or After Week 8 of the Treatment Period)
Description: Using the LogMAR score, lower values correspond to higher visual acuity. For example, a visual acuity of 20/20 corresponds to a LogMAR value of zero (0), and a visual acuity of 20/100 corresponds to a LogMAR value of 0.7.
Time Frame: At Week 12 or, if the Week 12 assessment is not available, at the last LogMAR assessment conducted at or after Week 8 of the Treatment Period
Population: The Intent-to-Treat (ITT) Population consisted of all randomized subjects who received any amount of study medication and had at least one evaluation of the primary efficacy variable (LogMAR score) at Week 8 or later and at Baseline.
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | IGIV-C 10% | Placebo
Number analyzed (Participants) | 29 | 24
LogMAR
  Baseline | 0.581 (0.209) | 0.533 (0.153)
  End of treatment (EOT) Week 12 or last assessment | 0.646 (0.309) | 0.557 (0.244)
  Change End of treatment (EOT) minus Baseline | 0.064 (0.220) | 0.024 (0.182)
Statistical Analysis 1: Comparison: IGIV-C 10% vs Placebo; The primary efficacy comparison for the change in LogMAR from baseline to endpoint was a two-way analysis of variance (ANOVA) with treatment group and center as fixed factors (main effect model); Test type: Superiority or Other; p = 0.49, ANOVA

2. Secondary Outcome: Proportion of Subjects Who Improve Visual Acuity From Baseline to Endpoint by ≥ 0.1 LogMAR
Time Frame: Last measurement at or later than Week 8
Population: Intent to Treat
Measure: Number; unit: percentage of participants
Arm/Group | IGIV-C 10% | Placebo
Number analyzed (Participants) | 29 | 24
percentage of participants | 24.1 | 20.8
Statistical Analysis 1: Comparison: IGIV-C 10% vs Placebo; Test type: Superiority or Other; p = 0.76, Cochran-Mantel-Haenszel — Adjusted for centers (including a Breslow-Day test for homogeneity of odd ratios across centers)

3. Secondary Outcome: Proportion of Subjects Who Improve Visual Acuity From Baseline to Endpoint by ≥ 0.2 LogMAR
Time Frame: Last measurement at or later than Week 8
Population: Intent to Treat
Measure: Number; unit: percentage of participants
Arm/Group | IGIV-C 10% | Placebo
Number analyzed (Participants) | 29 | 24
percentage of participants | 3.4 | 16.7
Statistical Analysis 1: Comparison: IGIV-C 10% vs Placebo; Test type: Superiority or Other; p = 0.13, Cochran-Mantel-Haenszel; Adjusted for centers (including a Breslow-Day test for homogeneity of odd ratios across centers)

4. Secondary Outcome: Mean Change in LogRAD Score From Baseline to Endpoint (RADNER Test)
Description: The RADNER test gives not only information about the subject's reading performance, but also about the reading speed (life quality) and the faults while reading. The RADNER reading charts (1, 2, and 3) contain sentences in paragraphs having a range of print sizes starting with the largest print at the top.The subject was randomly assigned one of the RADNER charts, and the charts were different between consecutive visits. The reading distance was 25 cm. The subject's score was corrected for reading speed and errors. The range of possible logRAD scores was from 2.0 (could not read the first paragraph) to -0.2, with higher scores indicating lower reading acuity and lower scores indicating higher reading acuity.
Time Frame: Last measurement at or later than Week 8
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: LogRAD
Arm/Group | IGIV-C 10% | Placebo
Number analyzed (Participants) | 29 | 24
LogRAD | 0.164 (0.343) | 0.159 (0.371)
Statistical Analysis 1: Comparison: IGIV-C 10% vs Placebo; Test type: Superiority or Other; p = 0.90, ANOVA; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.21 to 0.19]

5. Secondary Outcome: Proportion of Subjects With an Increase ≥ 2 or More Points in Lens Opacity Classification System (LOCS III) for Nuclear Opalescence, Nuclear Color, Cortical Cataract or Posterior Subcapsular Cataract Categories
Description: The LOCS III scale for cortical cataract and posterior subcapsular cataract opacity ranged from 1.0 to 5.0. The LOCS III scale for nuclear opalescence and for nuclear color was 1.0 to 6.0. For all scales, higher values indicate higher opacity, opalescence, or color.
Time Frame: Last measurement at or later than Week 8
Population: Intent to Treat subjects with cataract
Measure: Number; unit: participants
Arm/Group | IGIV-C 10% | Placebo
Number analyzed (Participants) | 19 | 15
participants | 0 | 0

6. Secondary Outcome: Presence of Fibrosis and Location Assessed by Slit-lamp
Time Frame: Last measurement at or later than Week 8
Population: Intent to Treat
Measure: Number; unit: participants
Arm/Group | IGIV-C 10% | Placebo
Number analyzed (Participants) | 29 | 24
participants | 1 | 3
Statistical Analysis 1: Comparison: IGIV-C 10% vs Placebo; Test type: Superiority or Other; p = 0.74, Cochran-Mantel-Haenszel; Adjusted to centers

7. Secondary Outcome: Mean Change From Baseline to Endpoint in Size of Lesion (Largest Dimension Relative to Disk Diameter) Assessed by Central Fluorescein Angiogram Reading Center
Time Frame: At end of treatment (12 weeks)
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: Disk Diameter
Arm/Group | IGIV-C 10% | Placebo
Number analyzed (Participants) | 29 | 24
Disk Diameter | 0.074 (0.209) | 0.173 (0.298)

ADVERSE EVENTS:
Arm/Group | IGIV-C 10% | Placebo
Serious Adverse Events (participants affected / at risk) | 1/30 | 5/27
Other Adverse Events (participants affected / at risk) | 21/30 | 15/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IGIV-C 10% (N=30) | Placebo (N=27)
Stent placement (Surgical and medical procedures) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abdominal pain, upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IGIV-C 10% (N=30) | Placebo (N=27)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Abdominal pain, upper (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Fatigue (General disorders) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 2 (2) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0)
Blood pressure increased (Investigations) | 2 (2) | 3 (3)
Blood urea increased (Investigations) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator must send a draft manuscript of the publication or abstract to the sponsor thirty days in advance of submission in order to obtain approval prior to submission of the final version for publication. This will be reviewed promptly and approval will not be withheld unreasonably. In case of a difference of opinion between the sponsor and the investigator(s), the contents of the publication will be discussed in order to find a solution which satisfies both parties.